CLINICAL TRIAL: NCT06068491
Title: Integrating Veteran-Centered Care for Advanced Liver Disease (I-VCALD)
Brief Title: Veteran-Centered Care for Advanced Liver Disease (Vet-CALD)
Acronym: Vet-CALD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: IIR 21-230; 1I01HX003541-01A1 (NIH)
Record Dates: First submitted 2023-09-28; First posted 2023-10-05 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Liver Diseases
Keywords: Patient-Centered Care; Randomized Controlled Trial; Delivery of Healthcare, Integrated
MeSH Terms: conditions — Liver Diseases

STUDY DESIGN:
Intervention Model Description: This is a hybrid type 1 effectiveness-implementation study utilizing formative implementation assessment prior to an effectiveness trial and assessment of implementation outcomes following the trial.
Who Masked: Outcomes Assessor
Masking Description: Data Collection Coordinator who conducts telephone surveys and chart reviews will be blinded to group assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1: Vet-CALD Intervention (Experimental): Vet-CALD Participants will receive the standard of care from their usual VA healthcare provider, plus they will participate in 5 monthly 60-minute care counselor sessions over a period of 6 months via VA Video Connect (VVC) or by telephone. The purpose of care counselor visits is to assess and cultivate the patient's understanding of their illness and identify personal healthcare goals. The counselor will be part of a centralized research care team (hepatologist and supportive care physician) and will work with each patient's usual VA care providers to help tailor treatment plans and education to better align with each patient's understanding of their disease prognosis and their healthcare goals and priorities.
  Interventions: Other: Vet-CALD
- Arm 2: Usual Care (No Intervention): Usual Care Participants will receive the standard of care from their usual VA healthcare provider. The care counselor will not contact the usual care condition participants.

INTERVENTIONS:
Other: Vet-CALD — Vet-CALD Participants will receive the standard of care from their usual VA healthcare provider, plus they will participate in 5 monthly 60-minute care counselor sessions over a period of 6 months via VA Video Connect (VVC) or by telephone. The purpose of care counselor visits is to assess and cultivate the patient's understanding of their illness and identify personal healthcare goals. The counselor will be part of a centralized research care team (hepatologist and supportive care physician) and will work with each patient's usual VA care providers to help tailor treatment plans and education to better align with each patient's understanding of their disease prognosis and their healthcare goals and priorities.
  Arms: Arm 1: Vet-CALD Intervention

SUMMARY:
Advanced liver disease is a serious illness that disproportionately affects Veterans, many of whom hope for curative liver transplantation. However, too few receive a transplant and most continue to suffer from increasing symptoms and hospitalizations. The proposed project uses a whole person, Veteran-centered approach that identifies Veterans with advanced liver disease using a population-based health management system and integrates curative and early supportive care using a telemedicine-based nurse care counselor to (1) discuss patient's understanding of illness severity and prognosis, (2) identify priorities and care preferences and (3) align curative and supportive care options to achieve patient priorities. Study outcomes include changes in (1) rates of consideration for liver transplantation, and (2) completion of serious illness discussions. Findings will inform adaptations to the intervention and facilitators for its dissemination.

DETAILED DESCRIPTION:
Project Background and Rationale: Advanced liver disease (AdvLD) is a serious illness. As many as half of AdvLD patients die within 2 years of developing liver complications, and nearly all suffer increasing symptoms and hospitalizations. Although many patients hope for curative liver transplantation, few receive it while experiencing an increasingly severe illness. In previous studies, many patients with AdvLD reported unmet curative and supportive care needs. They also reported preferences to align care with their outcome goals earlier in the AdvLD course than is now common. The Vet-CALD program is a Whole Health program in AdvLD that focuses on what matters most to patients, shared goals, and goal-aligned treatments, and could improve both curative and supportive care.

Project Objectives: The overall goal of the Vet-CALD project is to develop and test a novel sustainable Whole Health program in caring for patients with AdvLD. Using a hybrid type 1 effectiveness-implementation study design, the project will: (Aim 1) conduct a formative assessment of Vet-CALD implementation for Veterans with AdvLD; (Aim 2) evaluate the effectiveness of Vet-CALD in a randomized controlled study at 8 VA centers; and (Aim 3) conduct a summative assessment of implementation outcomes.

Project Methods: In Aim 1, the study team will conduct in-depth qualitative interviews with clinical stakeholders and patients to identify steps necessary to refine the Vet-CALD intervention, develop engagement processes for patients, and establish integrated workflows at the four targeted VA sites.

In Aim 2 the study team will conduct a randomized clinical trial (N=450) with patients from 8 VA medical centers assigned (1:1) to Usual Care vs. Vet-CALD Intervention. The Vet-CALD intervention will consist of a centralized research care counselor who will work with individual patients by telehealth (3 to 5 visits over 6 months) to assess and cultivate their understanding of their illness and identify personal healthcare goals. The counselor will be part of a centralized care team (hepatologist and supportive care physician) and will work with each patient's usual providers to help tailor treatment plans and education to better align with each patient's understanding of their disease prognosis and their healthcare goals and priorities.

In Aim 3, Summative assessment will provide context for the effectiveness results and inform necessary adaptations to and dissemination of Vet-CALD.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be between 18 and 80 years of age
* Patients must be Veterans
* Patients must have been in care at one of the recruiting sites with 1 or more encounters in primary care or GI/Hepatology in the last 24 months
* Patients must have advanced liver disease, defined by ICD-10 codes for cirrhosis complications (ever) or MELD 3.0 >12 or MELD-Na >12 or Fibroscan LSM >20kpa

Exclusion Criteria:

* Non-Veteran patients
* Patients who do not speak English, do not have access to a telephone or computers, or who are unable to complete a valid informed consent form after three attempts
* Patients who have already made significant progress toward our endpoints: a) with prior history of liver transplantation, or b) on the liver transplant waiting list, or c) had formal evaluation for liver transplantation in the past 3 years
* Patients with very limited life expectancy (advanced cancer, acute-on-chronic liver failure, and hospice patients)
* Patients hospitalized, or in long term facilities or nursing homes at the time they meet inclusion criteria
* Patients with chart diagnosis of uncontrolled mental health or schizophrenia

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
EHR documentation of consideration for liver transplantation change | 6 and 12 months
  Consideration of Liver Transplantation will be measured dichotomously by assigning a value of 1 if the patient's EHR includes at least one clinician note that documents consideration of liver transplantation as a potential treatment option for the patient within 6 months and 12 months of enrollment, and a value of 0 otherwise.
EHR documentation of goals of care conversation change | 6 and 12 months
  Goals of Care Conversation will be measured dichotomously by assigning a value of 1 if the patient's EHR includes at least one clinician note documenting discussion of goals of care planning within 6 months and 12 months of enrollment, and a value of 0 otherwise.

SECONDARY OUTCOMES:
Receipt of goal concordant care | 6 months
  Receipt of Goal Concordant Care will be measured using a 2-item survey. The first question defines patient preferences for either extending life or ensuring comfort. The second question assesses patients' perceptions of their current treatment with the same choices. The outcome is a dichotomous variable measuring whether preferences matched the patient's report of current care.
Health Related Quality of Life (HRQoL) | 6 months
  HRQoL will be measured at baseline and 6-months using the 10-item Patient-Reported Outcomes Measurement Information System (PROMIS) Global-10 instrument, which measures general domains of health including physical function, emotional distress, social health, as well as perceptions of general health that cut across domains, plus fatigue and pain. PROMIS-10 items are scored from 1 to 5 (Poor to Excellent; Not at All to Completely; Always to Never; Very Severe to None) and averaged to provide a mean HRQoL score ranging from 1 to 5. (T-score, higher score indicates better HRQoL.).
Perceived quality of shared decision-making | 6 months
  Perceived shared decision making will be measured using the 3-item CollaboRATE scale (scored 0 to 9; possible range 0-100; = 0.89 higher score indicates greater perceived shared decision-making and goal ascertainment)
Satisfaction with care | 6 months
  Satisfaction with Care will be measured using the 4-item Satisfaction with Care - Feeling Heard and Understood survey. (scored 0-4; Not at All True to Completely True; possible range 0-16; higher score indicates greater satisfaction with care and goal ascertainment).
Quality of symptomatic advanced liver disease (AdvLD) care | 12 months
  Quality of symptomatic care will be measured using a broad measure of quality based on selected AASLD's process-based quality indicators (QIs). Adherence to a given QI will be scored as 1 with evidence for satisfying the indicator. Quality of care at the patient level will be calculated by dividing the number of QIs for which that individual received the indicated care by the number of QIs for which the individual is eligible for during the 12-month follow up time.

CONTACTS AND LOCATIONS:
Overall Officials: Fasiha Kanwal, MD MSHS, Principal Investigator — Michael E. DeBakey VA Medical Center, Houston, TX; Anne M Walling, MD PhD, Principal Investigator — VA Greater Los Angeles Healthcare System, West Los Angeles, CA; Steven M. Asch, MD MPH, Principal Investigator — VA Palo Alto Health Care System, Palo Alto, CA
Locations (8):
- United States (8):
  - Central Arkansas Veterans Healthcare System , Little Rock, AR, Little Rock, Arkansas
  - VA Long Beach Healthcare System, Long Beach, CA, Long Beach, California
  - VA Palo Alto Health Care System, Palo Alto, CA, Palo Alto, California
  - VA Greater Los Angeles Healthcare System, West Los Angeles, CA, West Los Angeles, California
  - VA Connecticut Healthcare System West Haven Campus, West Haven, CT, West Haven, Connecticut
  - Miami VA Healthcare System, Miami, FL, Miami, Florida
  - VA North Texas Health Care System Dallas VA Medical Center, Dallas, TX, Dallas, Texas
  - Michael E. DeBakey VA Medical Center, Houston, TX, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
Data sharing will be accomplished through manuscript publications and presentations at scientific conferences. Requests for Limited Datasets (LDS) will be considered with appropriate data use agreements (DUAs) and IRB approvals. We will remove all HIPAA identifiers before sharing datasets. DUAs will limit use of the dataset and prohibit the recipient from identifying or re-identifying (or taking steps to identify or re-identify) any individual whose data are included in the dataset.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: starting 6 months after publication
Access Criteria: Aggregate data will be shared through manuscripts, reports and conference presentations. Corresponding Limited Data Sets (LDS) shared will include all the variables contained within our datasets (except for the 18 HIPAA identifiers). This will allow validation of our results by the recipients. Requests may be submitted to Fasiha Kanwal, MD, the overall PI, starting 6 months after publication and up to 4 years after the study ends.

REFERENCES:
- [Result] Kanwal F, Neuschwander-Tetri BA, Loomba R, Rinella ME. Metabolic dysfunction-associated steatotic liver disease: Update and impact of new nomenclature on the American Association for the Study of Liver Diseases practice guidance on nonalcoholic fatty liver disease. Hepatology. 2024 May 1;79(5):1212-1219. doi: 10.1097/HEP.0000000000000670. Epub 2023 Nov 9. PMID 38445559